CLINICAL TRIAL: NCT03142672
Title: Immediate Postoperative Pain and Recovery Time After Pulpotomy Performed Under General Anaesthesia in Young Children
Brief Title: Postoperative Pain and Recovery Time After Pulpotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SULTAN KELES, Assist. Prof.Dr., Aydin Adnan Menderes University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2016/764
Record Dates: First submitted 2017-04-26; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; child; pulpotomy; general anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Pulpotomy and tooth filling
  Interventions: Procedure: pulpotomy; Procedure: tooth filling
- Control group (Active Comparator): Tooth filling
  Interventions: Procedure: tooth filling

INTERVENTIONS:
Procedure: pulpotomy — vital endodontic procedure
  Arms: Experimental group
Procedure: tooth filling — tooth filling

SUMMARY:
The aim of this retrospective study was to compare immediate postoperative pain scores and the need for rescue analgesia in children who underwent pulpotomies and general restorative treatment and those who underwent general restorative treatment only, all under general anaesthesia.

DETAILED DESCRIPTION:
Ninety patients aged between 3 and 7 years who underwent full mouth dental rehabilitation under general anaesthesia were enrolled in the study and reviewed. The experimental group included patients who were treated with at least one pulpotomy, and the control group was treated with dental fillings only. The Wong-Baker FACES scale was used to evaluate self-reported pain and the need for rescue analgesia. The data were analysed using the Kruskal-Wallis test, two sample t- tests, chi-square tests and Pearson's correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent full mouth dental rehabilitation under GA because of their lack of chairside cooperation
* Patients with at least 1 pulpotomy were included in the experimental group (n=45), and patients treated with dental fillings only were included in the control group (n=45); a total of 90 patients were eligible for the study.

Exclusion Criteria:

* Children with special needs and those with any systematic problem (cardiac disease, diabetes, or intellectual disability) were excluded from the study.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Pain scores evaluation | An average of 1 year
  Wong Baker Faces Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Keles, Dr., Study Director — Pediatric dentistry

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jensen B. Post-operative pain and pain management in children after dental extractions under general anaesthesia. Eur Arch Paediatr Dent. 2012 Jun;13(3):119-25. doi: 10.1007/BF03262857. PMID 22652208